CLINICAL TRIAL: NCT06784323
Title: A Culturally Tailored Anti-inflammatory Diet for American Patients With Ulcerative Colitis
Brief Title: Tailored Anti-Inflammatory (A-I) Diet for Americans With Ulcerative Colitis (UC)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Oriana Mazorra Damas, Associate Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20240857; 1R01DK140964-01 (NIH)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catered diet group (Experimental): Participants will be in this arm for up to 8 weeks.
  Interventions: Behavioral: Catered diet; Behavioral: Diet guidance sessions; Behavioral: Dietary counseling; Behavioral: Feedback sessions
- Diet guidance sessions group (Experimental): Participants will be in this arm for up to 8 weeks.
  Interventions: Behavioral: Catered diet; Behavioral: Diet guidance sessions; Behavioral: Dietary counseling; Behavioral: Feedback sessions

INTERVENTIONS:
Behavioral: Catered diet — For a period of 8 weeks the participant will receive catered food, the study team will provide the participants breakfast, lunch and dinner. Participants will receive catered food for 3 daily meals, and record daily food intake. Catered diet will be sent to participants' homes on a weekly basis. The diet will consist of primarily whole foods with few additives, with a focus on American staple foods.
Behavioral: Diet guidance sessions — Participants will receive virtual weekly diet guidance with a dietitian regarding food safety preparation methods and cooking practices. Patients will receive weekly gift cards for grocery stipend. On average, initial counseling session with dietitian will last 30 minutes, and 7 follow-up sessions will last 20 minutes.
Behavioral: Dietary counseling — Participants will receive dietary counseling weekly on Zoom for up to 30 minutes. Dietitian will meet with participants to explain benefits of adhering to diet therapy.
Behavioral: Feedback sessions — Participants will be involved in one-time 50-minute feedback session over Zoom with dietitian and principal investigator. During the session, participants will discuss preferred foods/recipes during active disease, likeability of recipes, ease of recipe preparation, dietary adherence, and healthy food affordability.

SUMMARY:
The purpose of this study is to test the effect of an anti-inflammatory diet that incorporates native foods of the American diet on disease remission in American patients with Ulcerative Colitis (UC) and to identify biomarkers of response to dietary therapy.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis with ulcerative colitis from medical records.
* Self-Identify as American
* Ages 16-75
* SCCAI between 3-9 (no greater than 12 bowel movements a day)
* Fecal calprotectin > 150mg/dl.
* On stable medications for their disease for the past 3 months
* Likeability of American foods (sandwiches, BBQ or grilled meats and vegetables, baked potatoes, smoothies, salmon, oatmeal, avocado, soups)
* No recent Inflammatory Bowel Disease (IBD) related hospitalization in the last month.

Exclusion Criteria:

* Diagnosis of Crohn's Disease (CD).
* Prior ileoanal anastomosis (J-pouch) or diversion
* No recent hospitalizations on the last 4 weeks
* No Clostridium difficile or enteric infections on the last 4 weeks
* No use of probiotics on the last 4 weeks
* Patients following the specific carbohydrate diet or mediterranean diet or anti-inflammatory diet
* No active cancer or conditions limiting their ability to follow a diet (heart failure, end stage renal disease)
* Pregnancy, breastfeeding or planning to become pregnant during study period
* Use of Total Parenteral Nutrition at the time of screening and during the study period
* Other significant or life-threatening co-morbidities
* The need for antibiotic use during the study period
* Adults unable to consent
* Ages less than 16 and > 75 years old
* Prisoners

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical remission after diet intervention measured by simple clinical colitis activity index (SCCAI) | Up to 8 weeks
  Will be measured with SCCAI <=2.0. Score of 2 or less indicates remission from ulcerative colitis (UC).
Fecal calprotectin | Up to 8 weeks
  Will be measured <150 μg/g

CONTACTS AND LOCATIONS:
Overall Officials: Oriana Damas, MD, MSCTI, Principal Investigator — University of Miami Health System
Locations (1):
- University of Miami Health System, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No